CLINICAL TRIAL: NCT03713775
Title: Weight Loss in Elderly Patients With Atrial Fibrillation (LOSE-AF): A Randomised Controlled Trial
Brief Title: LOSE-AF: Can Weight Loss Help Patients With Atrial Fibrillation?
Acronym: LOSE-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID13511-SP001-AC002; 242939 (Other: IRAS)
Record Dates: First submitted 2018-10-15; First posted 2018-10-22 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation; Overweight and Obesity
MeSH Terms: conditions — Atrial Fibrillation; Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is an open-label randomised controlled study and patients will be aware of their treatment allocation. Potentially subjective measurements will be undertaken by observers blinded to treatment allocation; in particular, all imaging and ECG monitoring data will be anonymised prior to post-processing, and PPT score will be assessed by a research nurse blinded to treatment allocation. All study assessments will be coded and recorded blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meal Replacement Weight Loss Programme (Experimental): The study intervention will be the referral to a commercial provider (CP) offering a Meal Replacement Weight Loss Programme with behavioural support. Briefly, participants will be referred to a nominated CP local counsellor who will set regular appointments during a period of 32-to-36 weeks to provide behavioural support, weight monitoring, and deliver formula meals. All counsellors delivering the programme will receive, beyond their routine training and accreditation, specific information related to this study before being allocated patients. The programme conventionally includes the 3 phases (meal replacement phase, transition phase, and weight maintenance phase) but the Consultant will have full discretion to modify and tailor this programme to suit each individual participant.
  Interventions: Other: Meal Replacement Weight Loss Programme
- Usual Care (Active Comparator): Participants randomised to the control group will receive best usual care, consisting of a one-off face-to-face consultation on weight loss with a nurse at baseline (~15 min at the John Radcliffe Hospital, Oxford) together with supporting written information (i.e. a copy of the booklet 'Facts not fads - Your simple guide to healthy weight loss.')
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Meal Replacement Weight Loss Programme — The study intervention will be the referral to a commercial provider (CP) offering a Meal Replacement Programme. Briefly, participants will be referred to a nominated CP local counsellor who will set regular appointments during a period of 32-to-36 weeks to provide behavioural support, weight monitoring, and deliver formula meals. All counselors delivering the programme will receive, beyond their routine training and accreditation, specific information related to this study before being allocated patients.
  Arms: Meal Replacement Weight Loss Programme
Other: Usual Care — Participants randomised to the control group will receive best usual care, consisting of a one-off face-to-face consultation on weight loss with a nurse at baseline (~15 min), together with supporting written information.
  Arms: Usual Care

SUMMARY:
Background Atrial fibrillation (AF) affects over 1 million individuals in the UK and results in costs of over £450 million per year to the National Health Service (NHS). Current rhythm control strategies are limited by high recurrences of AF. New strategies tackling more upstream pathophysiological mechanisms are most needed. The incidence and prevalence of AF markedly increase with age, whilst obesity is the strongest modifiable risk factor for AF. Preliminary data in relatively young patients suggest that weight loss programmes may reduce AF burden and improve AF-related symptoms. Such programmes could be a widely-applicable and cost-effective option in AF management if they are also effective in elderly patients with AF, particularly if they also improve physical performance.

Aim The aim of this study is to investigate whether, in older overweight/obese AF patients, referral to a weight loss programme with meal replacement & behavioral support can reduce AF-recurrences and improve physical performance compared to usual care.

Study design Parallel-group, open-label, multi-centre randomised controlled trial. Elderly individuals (60-85 years) with persistent AF and elevated body mass index (BMI; ≥ 27 kg/m2) will be recruited. Participants will be randomly allocated (1:1) to (a) referral to a meal replacement programme with behavioral support (intervention) or (b) usual care (control) for 32-to-36 weeks. The primary endpoints are AF recurrence and physical performance test (PPT) score. Participants randomised to the study intervention will be referred to a commercial provider (CP) providing the intervention. The co-primary endpoints of AF recurrence & PPT score will be analysed irrespective of compliance during the scheduled treatment period following an intention-to-treat principle.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained arrhythmia, and is associated with a two-fold increase in the risk of premature death. Morbidity and mortality related to stroke, heart failure, myocardial infarction, and reduced quality of life, are all common in patients with AF. AF therefore represents a burgeoning public health problem, affecting over 1 million patients in the UK and resulting in estimated costs of over £450 million per annum. The main drivers of AF-related costs are hospitalizations (over £270 million for admissions annually) and outpatient encounters (approximately £50 million for General Practitioner consultations and £36 million for specialist clinic referrals annually)11. Recurrence of AF remains a clinical challenge despite pharmacological and interventional rhythm control strategies. Moreover, currently available therapies have not been consistently shown to reduce AF recurrence and the risk of major adverse events, or to improve long-term prognosis.

The incidence and prevalence of AF are closely linked to increasing age and excess weight. On one hand, advanced age is the most important non-modifiable risk factor for AF and the corollary is that AF is associated with frailty and impaired physical function. Meanwhile, excess weight is of particular interest as results from four large community-based European studies clearly demonstrated that elevated body mass index (BMI) is the strongest modifiable risk factor for incident AF. A large-scale observational cohort study reported a 4% increase in AF-risk per 1-unit increase in body mass index (BMI) after adjustment for cardiovascular risk factors and interim myocardial infarction or heart failure. Moreover, a recent Mendelian randomization study confirmed a causal relationship between increased BMI and incident AF. The precise mechanisms by which obesity increases the risk of development and maintenance of AF are incompletely understood; potential contributors include left atrial (LA) enlargement, left ventricular (LV) hypertrophy, diastolic dysfunction, altered cardiac energetics, and inflammatory/oxidative signalling from the epicardial adipose tissue.

Very low calorie diets, providing less than 800 kcal/d have been used for many years as highly effective methods for inducing weight loss, leading to consistent reductions in visceral fat and overall adiposity. A systematic review showed weight loss at 1 year of 8-14 kg, which was 4.3 kg (95% CI: 1.1 kg, 7.4 kg) greater than the comparator interventions. The historical limitation of very low calorie diets has historically been long-term effectiveness, and there has been growing interest in the use of total meal replacement sachets as part of a wider behavioural programme. This includes individualised one-to-one counselling to motivate and encourage adherence to the diet, as well as support to establish a healthy eating plan when individuals reintroduce food. Results from DiRECT (a cluster-randomised trial assessing a meal replacement programme in patients with type II diabetes) were published recently in The Lancet: the intervention arm reached an average weight loss of 10 kg at 1 year with 45% of individuals achieving complete remission of type II diabetes, which is also a relevant risk factor for AF. Preliminary data suggest that such a programme proved highly effective in reducing AF symptoms in a relatively young group of AF patients where the diet resulted in significant weight loss (>10kg) sustained to 15 months. However, it remains unclear whether the beneficial effects of weight loss translate in (a) reducing AF recurrences and (b) whether they also extend to the more typical elderly patient population with AF, as reversing cardiac remodelling may prove more difficult in aged hearts. Additionally, the balance between beneficial and detrimental effects of weight loss in the elderly may be dependent on preservation of muscle strength.

The aim of this study is to investigate whether, in older overweight/obese AF patients, referral to a weight loss programme with meal replacement & behavioral support can reduce AF-recurrences and improve physical performance compared to usual care.

This is a parallel-group, open-label, randomized controlled study to determine whether substantial weight reduction through referral to a weight loss programme with meal replacement & behavioral support in older patients who are overweight/obese with persistent AF can reduce AF recurrences and symptoms and improve the adverse cardiometabolic profile and physical performance. The expected duration of such programme is approximately 8 months, with a total of two study visits (at baseline and at 8 months). AF-related symptoms (primary endpoint) are assessed at baseline and at approximately 8 months after the commencement of the intervention using the AFSS symptom score.

Elderly individuals (60-85 years) with elevated BMI (≥27 kg/m2), who are scheduled for a DCCV with a diagnosis of persistent AF will be recruited. Participants will be randomised (1:1) to (a) weight loss programme for a total of ~8 months (intervention) or (b) usual care; i.e., nurse-based consultation and supporting written material (control). All participants will undergo a baseline visit (prior to randomisation) and a follow-up visit at ~8 months. Both study visits will include a physical performance test (PPT), AF symptom assessment using the AFSS score, anthropometric measurements, quality of life assessment, Patient Health-Resource Use Questionnaire (PRUQ), MR scan, and blood sample collection. Additionally, prolonged ECG monitoring, and patient reported outcome measures (PROMs) will also be acquired at the 8-month visit. Finally, at approximately 4 months patients will be asked to complete interim questionnaires (including PRUQ, PROMs, Quality of Life) by post/telephone.

In the LOSE-AF trial, the intervention is at very low risk of adverse events and no Trial Steering Committee or Clinical Trial Authorization is required. The study will be coordinated by the Trial Management Committee (TMC), consisting of at least one core study investigator (a medically qualified clinician), and the research nurse. The TMC will be responsible for the day-to-day management of the trial and will meet regularly.

ELIGIBILITY:
Inclusion Criteria:

* Persistent AF
* Body mass index ≥27 kg/m2

Exclusion Criteria:

* Planned catheter ablation for AF within 8 months
* Learning difficulties or unable to understand English
* Participation in another research trial involving an investigational product or weight loss programme in the prior 3 months
* Current treatment with anti-obesity drugs
* Uncontrolled endocrine disorders
* Diabetes requiring insulin
* Active gout or history of recurrent gout
* Ongoing gallbladder disease
* Serious underlying medical or psychiatric disorder; e.g., known cancer or any other significant disease affecting short-term life expectancy; severe valvular disease, myocardial infarction or stroke within the previous 6 months; severe heart failure; eating disorder or purging behaviour; severe psychotic disorder requiring hospitalisation or supervised care, active liver disease (except non-alcoholic fatty liver disease).
* Unintentional weight loss of more than 5 kg within the prior 6 months
* Gastrointestinal malabsorption
* Unstable INR (persistently <2 for >14 days) or supra-therapeutic levels with concomitant bleeding or requiring hospitalisation
* Substance abuse
* Taking varenicline (smoking cessation medication)
* Chronic renal failure of stage 4 or 5
* Porphyria

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation symptoms severity (0-35) | 8 months
  Toronto AF Severity Scale (AFSS) score (points) - This is a validated questionnaire assessing AF symptom severity (range, 0 no symptoms to 35 severe symptomatology).
  Reference: Dorian P, Jung W, Newman D, et al. The impairment of health-related quality of life in patients with intermittent atrial fibrillation: implications for the assessment of investigational therapy. J Am Coll Cardiol 2000;36:1303-9.

SECONDARY OUTCOMES:
Atrial fibrillation burden | 8 months
  The burden (proportion) of atrial fibrillation (AF) during a 14-day ECG monitoring period using a wearable patch (AF is diagnosed and categorised according to the accepted definition based on ECG morphology including absence of p waves, irregularly irregular RR intervals, absence of isoelectric baseline, and/or presence of fibrillatory waves)
Atrial fibrillation symptoms burden (3.25-30) | 4 & 8 months
  Toronto AF Severity Scale (AFSS) score (points) - This is a validated questionnaire encompassing 12-item AF-specific scale, assessing AF symptom burden (range, 3.25 minimally symptomatic episode to 30 highly symptomatic episode) and AF symptom severity (range, 0 no symptoms to 35 severe symptomatology).
  Reference: Dorian P, Jung W, Newman D, et al. The impairment of health-related quality of life in patients with intermittent atrial fibrillation: implications for the assessment of investigational therapy. J Am Coll Cardiol 2000;36:1303-9.
Atrial fibrillation symptoms severity (0-35) | 4 months
  Toronto AF Severity Scale (AFSS) score (points) - This is a validated questionnaire encompassing 12-item AF-specific scale, assessing AF symptom burden (range, 3.25 minimally symptomatic episode to 30 highly symptomatic episode) and AF symptom severity (range, 0 no symptoms to 35 severe symptomatology).
  Reference: Dorian P, Jung W, Newman D, et al. The impairment of health-related quality of life in patients with intermittent atrial fibrillation: implications for the assessment of investigational therapy. J Am Coll Cardiol 2000;36:1303-9.
Quality of Life (QoL) by EuroQoL EQ-5D-5L utility score | 4 & 8 months
  EuroQoL EQ-5D-5L utility score (points)
Patient Reported Outcome Measures (PROMs) | 4 & 8 months
  Questionnaire to assess adherence and feedback on the weight loss method qualitatively
Patient Resource Use Questionnaire (PRUQ) | 4 & 8 months
  Questionnaire (points)
Body mass | 8 months
  Body Weight by weighing scales (kg)
Body composition profile | 8 months
  Total fat (ml) by MRI (Dixon-sequence)
Body composition profile: visceral fat | 8 months
  Visceral fat (ml) by MRI (Dixon-sequence)
Body composition profile: skeletal muscle | 8 months
  Skeletal muscle volumes (ml) by MRI (Dixon-sequence)
Skeletal muscle energetics (quadriceps femoris) | 8 months
  Phosphocreatine (PCr) recovery rate (sec) by 31P magnetic resonance spectroscopy (31P-MRS)
Left ventricular (LV) energetics | 8 months
  LV PCr/ATP ratio by 31P-MRS
Left Ventricular (LV) structure | 8 months
  LV volumes (ml) by cardiac MRI
Left Atrial (LA) structure | 8 months
  LA volumes (ml) by cardiac MRI
Left Ventricular (LV) function | 8 months
  LV function (%) by cardiac MRI
Left Atrial (LA) function | 8 months
  LA function (%) by cardiac MRI
Left Atrial (LA) Flow | 8 months
  LA blood flow (% of stasis) by cardiac MRI
Left Ventricular (LV) Flow | 8 months
  LV blood flow (residual volume %) by cardiac MRI
Health economics outcomes | through study completion, an average of 2 year
  Incremental Cost-Effectiveness Ratio (Cost per Quality-Adjusted Life Year)
Physical Performance Test (PPT) score (points) | 8 months
  The modified Physical Performance Test (PPT) is derived by evaluating performance in daily activities, with 36 being the best total score for the test. The overall PPT score (co-primary outcome) is derived from performance undertaking six standardized tasks that are timed (walking ~15 m, putting on and removing a coat, picking up a penny ~30 cm in front of the dominant side foot, standing up from a ~40 cm chair, lifting a ~3 kg book to a shelf ~30 cm above shoulder height, climbing one flight of 10 stairs), plus 3 additional tasks (performing a progressive Romberg test with feet side-by-side, semi-tandem and full-tandem, climbing up and down four flights of 10 stairs, and performing a 360-degree turn).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Casadei, MD DPhil, Principal Investigator — University of Oxford
Locations (1):
- Oxford Centre for Magnetic Resonance (OCMR), Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No